CLINICAL TRIAL: NCT07075471
Title: Real-World Patient Experience of Vimseltinib for the Treatment of Tenosynovial Giant Cell Tumor
Brief Title: Tenosynovial Giant Cell Tumor (TGCT) Real-World Participant Experience With Vimseltinib
Status: Recruiting | Type: Observational
Sponsor: Deciphera Pharmaceuticals, LLC (Industry)
Responsible Party: Sponsor
Other Study IDs: DCC-3014-04-001
Record Dates: First submitted 2025-07-11; First posted 2025-07-20 (Actual); Last update posted 2025-11-05 (Actual); Status verified 2025-11

CONDITIONS: Tenosynovial Giant Cell Tumor
MeSH Terms: conditions — Giant Cell Tumor of Tendon Sheath

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 12 Months
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
The goal of this observational study is to better understand real-world use of vimseltinib, treatment patterns, and health-related quality of life in participants treated with vimseltinib for TGCT.

This study will collect data in an observational disease registry involving no intervention to the participants and will not influence standard medical care or impact treatment decisions for participants.

ELIGIBILITY:
Inclusion Criteria:

1. Diagnosis of TGCT according to medical records
2. Prescribed vimseltinib per the approved label requirements. Participants are eligible if either (A) the decision to receive vimseltinib has been made but treatment has not yet been initiated or (B) the decision to receive vimseltinib has been made and participant has received first dose of prescribed vimseltinib less than 6 months prior to study enrollment
3. Has provided informed consent and medical records release

Exclusion Criteria:

1. Participant has received any other systemic agent for the treatment of TGCT during the 6 months prior to starting treatment with vimseltinib
2. Participant has received the first dose of prescribed vimseltinib in the current treatment course more than 6 months before study enrollment
3. Participant is active in an interventional clinical trial of vimseltinib

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Participants being treated for TGCT with vimseltinib in the community setting.
Sampling Method: Non-Probability Sample
Enrollment: 100 (Estimated)
Dates: Start 2025-09-03 (Actual); Primary Completion 2027-09 (Estimated); Study Completion 2027-09 (Estimated)

PRIMARY OUTCOMES:
Duration of Vimseltinib Treatment | Baseline up to 12 months
Time to Discontinuation of Vimseltinib | Baseline to Discontinuation (Estimated up to 12 months)

CONTACTS AND LOCATIONS:
Overall Officials: Clinical Team, Study Director — Deciphera Pharmaceuticals, LLC
Locations (1):
- Synexus Clinical Research, US INC, Wilmington, North Carolina, United States

IPD SHARING:
Plan to Share IPD: No